CLINICAL TRIAL: NCT00350870
Title: Maximizing the Efficacy of Cognitive Behavioral Therapy With Medication and Contingency Management
Brief Title: CBT With Disulfiram and Contingency Management
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0408026992; 5R01DA019078 (NIH)
Record Dates: First submitted 2006-07-07; First posted 2006-07-11 (Estimated); Results first posted 2014-12-03 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2014-11

CONDITIONS: Cocaine Abuse
Keywords: disulfiram; cognitive behavioral therapy; contingency management; drug abuse therapy; educational/resource design/development
MeSH Terms: conditions — Cocaine-Related Disorders | interventions — Disulfiram

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Placebo (Placebo Comparator): Placebo (plus Cognitive Behavioral Therapy- CBT)
  Interventions: Drug: Placebo
- Disulfiram (Active Comparator): Disulfiram (plus CBT)
  Interventions: Drug: disulfiram
- Placebo plus Contingency Management (Placebo Comparator): Placebo plus Contingency Management for cocaine abstinence and medication compliance (in addition to CBT).
  Interventions: Behavioral: Placebo plus Contingency Management
- Disulfiram plus Contingency Management (Active Comparator): Disulfiram plus Contingency Management for cocaine abstinence and medication compliance (in addition to CBT).
  Interventions: Drug: Disulfiram plus Contingency Management

INTERVENTIONS:
Drug: disulfiram — 250mg per day of Disulfiram plus CBT
  Other Names: antabuse; antabus
  Arms: Disulfiram
Drug: Placebo — Placebo plus CBT
  Arms: Placebo
Behavioral: Placebo plus Contingency Management — Placebo plus Contingency Management for cocaine abstinence and medication compliance in addition to CBT
  Arms: Placebo plus Contingency Management
Drug: Disulfiram plus Contingency Management — 250mg of Disulfiram plus Contingency Management for cocaine abstinence and medication compliance plus CBT.
  Other Names: antabuse; antabus
  Arms: Disulfiram plus Contingency Management

SUMMARY:
This is a study of four treatments for chronic cocaine use and may help study participants to control their drug use. All participants will receive weekly individual cognitive behavioral therapy (CBT).

DETAILED DESCRIPTION:
This study will compare four types of treatment involving skills training and incentives for attending sessions or taking study medication. Disulfiram is a widely prescribed deterrent to alcohol use. In addition to weekly cognitive behavioral therapy (CBT), participants will be assigned to one of the following treatments:

1. placebo
2. disulfiram
3. placebo plus incentives for cocaine abstinence and medication compliance (prize CM)
4. disulfiram plus incentives for cocaine abstinence and medication compliance

ELIGIBILITY:
Inclusion Criteria:

* 18-50 year old
* cocaine dependent
* willing to sign consent
* willing to accept randomization to intervention

Exclusion Criteria:

* significant medical conditions
* psychiatric disorder with current use of prescribed psychotropic medication
* lifetime schizophrenia or bipolar disorder
* suicidality or homicidality
* unlikely to be able to complete 1 year follow up
* unable to speak or read English at a third grade level

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 181 (Actual)
Dates: Start 2005-04; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen M. Carroll, PhD, Principal Investigator — Yale University
Locations (1):
- APT Foundation, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Worhunsky PD, Stevens MC, Carroll KM, Rounsaville BJ, Calhoun VD, Pearlson GD, Potenza MN. Functional brain networks associated with cognitive control, cocaine dependence, and treatment outcome. Psychol Addict Behav. 2013 Jun;27(2):477-88. doi: 10.1037/a0029092. Epub 2012 Jul 9. PMID 22775772
- [Derived] Carroll KM, Nich C, Shi JM, Eagan D, Ball SA. Efficacy of disulfiram and Twelve Step Facilitation in cocaine-dependent individuals maintained on methadone: a randomized placebo-controlled trial. Drug Alcohol Depend. 2012 Nov 1;126(1-2):224-31. doi: 10.1016/j.drugalcdep.2012.05.019. Epub 2012 Jun 12. PMID 22695473

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 181 patients were assessed for eligibility. 40 were found to be ineligible, and 42 did not complete the screening. 99 were randomized, but only 80 started (defined as having at least 1 day of study medication).
Period: Overall Study
Arm/Group | Placebo | Disulfiram | Placebo Plus Contingency Management | Disulfiram Plus Contingency Management
Started | 27 | 28 | 22 | 22
Had at Least 1 Day of Med | 19 | 24 | 18 | 19
Completed | 5 | 11 | 6 | 7
Not Completed | 22 | 17 | 16 | 15
Not completed — Withdrawal by Subject | 21 | 17 | 15 | 14
Not completed — Physician Decision | 1 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Disulfiram | Placebo Plus Contingency Management | Disulfiram Plus Contingency Management | Total
Number analyzed (Participants) | 27 | 28 | 22 | 22 | 99
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.6 (8.8) | 39.8 (7.5) | 38.5 (7.4) | 39.3 (6.3) | 39.3 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 9 | 7 | 7 | 27
  Male | 23 | 19 | 15 | 15 | 72
Race/Ethnicity, Customized [Number; unit: participants]
  Cuacasian | 12 | 11 | 3 | 13 | 39
  African-American | 12 | 14 | 15 | 8 | 49
  Latino | 2 | 3 | 2 | 0 | 7
  Multiracial/Other | 1 | 0 | 2 | 1 | 4

OUTCOME MEASURES:

1. Primary Outcome: Change in Cocaine Use by Self Report
Description: Self-reports of substance use will be documented at each contact via the Substance Use Calendar. Similar to the Form-90 and the Time Line Follow-Back, which have been shown to be reliable and valid instruments for monitoring substance use and other outcomes in longitudinal studies202-204, the Substance Use Calendar allows a flexible, continuous evaluation of substance use on a daily basis.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of days abstinent
Arm/Group | Placebo | Disulfiram | Placebo Plus Contingency Management | Disulfiram Plus Contingency Management
Number analyzed (Participants) | 27 | 28 | 22 | 22
percentage of days abstinent | 72.2 (27.3) | 79.2 (18.1) | 91.1 (13.6) | 69.6 (31.7)

2. Primary Outcome: Change in Cocaine Use by Urine Toxicology Results
Description: We will use the Roche onsite TESTCUP system for detection of cocaine, methamphetamine, THC, benzodiazepenes, and opioids.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: percentage of negative urines
Arm/Group | Placebo | Disulfiram | Placebo Plus Contingency Management | Disulfiram Plus Contingency Management
Number analyzed (Participants) | 27 | 28 | 22 | 22
percentage of negative urines | 17.9 (32.3) | 30.1 (39.6) | 53 (41) | 42.6 (43.7)

ADVERSE EVENTS:
Arm/Group | Placebo | Disulfiram | Placebo Plus Contingency Management | Disulfiram Plus Contingency Management
Serious Adverse Events (participants affected / at risk) | 10/27 | 10/28 | 7/22 | 7/22
Other Adverse Events (participants affected / at risk) | 12/27 | 17/28 | 10/22 | 17/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Disulfiram (N=28) | Placebo Plus Contingency Management (N=22) | Disulfiram Plus Contingency Management (N=22)
Medical Hospitilization (Surgical and medical procedures) | 2 (2) | 1 (1) | 2 (2) | 2 (3)
Substance Use Hospitalization (General disorders) | 6 (8) | 8 (9) | 4 (4) | 5 (7)
Psychiatric Hospitalization (Psychiatric disorders) | 2 (2) | 1 (1) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=27) | Disulfiram (N=28) | Placebo Plus Contingency Management (N=22) | Disulfiram Plus Contingency Management (N=22)
Drowsiness (General disorders) | 2 (2) | 5 (5) | 2 (2) | 2 (2)
Fatigue (General disorders) | 1 (1) | 3 (3) | 2 (2) | 3 (3)
Restlessness (General disorders) | 2 (2) | 4 (4) | 1 (1) | 3 (3)
Headache (General disorders) | 4 (4) | 5 (5) | 1 (1) | 6 (6)
Tremors (General disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Optic Neuritis (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Nausea and Vomiting (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1) | 4 (4)
Diarrhea/Constipation (Gastrointestinal disorders) | 2 (2) | 4 (4) | 1 (1) | 5 (5)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Aftertaste (General disorders) | 1 (1) | 7 (7) | 2 (2) | 7 (7)
Peripheral Neuritis (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes